CLINICAL TRIAL: NCT07379008
Title: Safety and Efficacy of a Non-Setting Paste in Bone Defect Reconstruction
Brief Title: Safety and Efficacy of Non-Setting Paste in Bone Defect Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biovico Sp. z o.o. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2.0 25.01.2024
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Bone Diseases; Bone Cysts; Bone Neoplasm; Enchondromatosis; Bone Defects
Keywords: Bone substitute; Bone defect reconstruction; Benign bone tumor; Bone regeneration; Osteoconductivity; Injectable bone graft; Bone remodeling
MeSH Terms: conditions — Bone Diseases; Bone Cysts; Bone Neoplasms; Enchondromatosis

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized, unblinded, single-arm clinical trial without a control group, focusing on safety and efficacy evaluation of the bone substitute material.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): A total of 29 patients, aged 18 to 75, who required bone defect filling following curettage of benign bone tumors or tumor-like lesions, underwent surgical implantation of a non-setting bone substitute paste to fill the resulting defects.
  Interventions: Device: Non-setting paste

INTERVENTIONS:
Device: Non-setting paste — Non-setting paste is injected into bone defects during surgical procedures for bone void reconstruction.

SUMMARY:
This study aims to evaluate the safety and efficacy of a novel bone substitute material for the treatment of bone defects in patients requiring defect filling following the excision of benign bone tumors, cysts, or similar lesions.

A total of 29 patients will undergo surgical intervention during which the bone substitute paste is applied to the defect site. Patients will be followed for 12 months, with radiographic assessments to monitor bone healing. The primary objectives of the study are to assess the adequacy of bone regeneration and to evaluate the safety profile of the material.

DETAILED DESCRIPTION:
This prospective, non-randomized, unblinded clinical trial evaluates a non-setting paste for bone defect reconstruction. The study is conducted at two centers in Poland (Gdańsk and Zgorzelec).

The study enrolls 29 patients aged 18-75 years who require bone defect filling following curettage of benign bone tumors and tumor-like lesions (cysts, chondromas, enchondromas). Patients with inflammatory conditions, autoimmune diseases, hypersensitivity to any components, or those using medications affecting bone remodeling are excluded.

Bone remodeling is assessed radiologically at 6 weeks, 6 months, and 12 months using the modified four-grade Neer classification. Success is defined as achieving Grade I (>75% remodeling) or Grade II (51-75% remodeling) at 12 months. Secondary endpoints include safety monitoring and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Qualified for bone defect filling procedures of various origins (e.g., bone void reconstruction following curettage of benign bone tumors, cysts, chondromas)
* Age 18 to 75 years
* Signed informed consent form

Exclusion Criteria:

* Acute or chronic inflammatory conditions in the surgical area
* Systemic inflammatory and autoimmune diseases
* Severe degenerative diseases
* Confirmed hypersensitivity to product components
* Skin inflammation or dermatological disease at the surgical site
* Use of medications that may affect bone remodeling (e.g., bisphosphonates)
* Use of corticosteroid-based medications
* Participation in another clinical trial
* Pregnancy or breastfeeding status

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2025-11-12 (Actual); Study Completion 2025-11-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of Non-setting Paste in Bone Defect Remodeling at 12 Months | 12 months post-surgery
  Success is defined as achieving Grade I (>75% bone remodeling with >75% material resorption) or Grade II (51-75% bone remodeling with 51-75% material resorption) according to the modified four-grade Neer classification system, assessed by radiographic examination with independent expert review.

SECONDARY OUTCOMES:
Safety profile assessment | Throughout 12-month study period
  Comprehensive monitoring of adverse events (AEs) and serious adverse events (SAEs) using the MedDRA classification system.
Bone remodeling progression at 6 weeks and 6 months | 6 weeks, 6 months post-implantation
  Assessment using modified Neer classification (Grade I-IV) by radiographic examination at 6 weeks and 6 months post-surgery to evaluate the progression of bone healing over time.
Patient Satisfaction | 12 months post-surgery
  Evaluation of patient satisfaction with clinical trial participation and treatment outcomes using structured questionnaires.
Treatment discontinuation rate | Throughout 12-month study period
  Number and percentage of patients who discontinue treatment due to device-related adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopaedics and Traumatology, Medical University of Gdansk, Gdansk, Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No